CLINICAL TRIAL: NCT05155904
Title: In-hospital Mortality of Patients With Veno Arterial ECMO: a Prospective Observational Study
Brief Title: Outcomes of Veno Arterial ECMO
Acronym: ECMOCARD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_204
Record Dates: First submitted 2021-11-16; First posted 2021-12-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mortality; Extra Corporeal Membrane Oxygenation
Keywords: veno arterial; mortality; extra corporeal membrane oxygenation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
veno arterial (VA) extra corporeal membrane oxygenation (ECMO) is a rescue therapy with various indications including refractory cardiac arrest and refractory cardiogenic shock. Amiens hospital university has an ECMO program and is a regional center to address patients requiring VA ECMO. In spite of the application of international guidelines, the mortality of patients with VA remains high with an admitted survival rate at hospital discharge at 40%.

ELIGIBILITY:
Inclusion Criteria:

* age : ≥ 18
* Patient with a VA ECMO

Exclusion Criteria:

* age<18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in Amiens hospital university beneficing of a veno arterial (VA) extra corporeal membrane oxygenation (ECMO).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Up to hospital discharge, an average of 1 month
  In-hospital mortality of patients with : veno arterial (VA) extra corporeal membrane oxygenation (ECMO)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No